CLINICAL TRIAL: NCT02937272
Title: A Phase 1 Study of LY3200882 in Patients With Solid Tumors
Brief Title: A Study of LY3200882 in Participants With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16185; I8X-MC-JECA (Other: Eli Lilly and Company); 2016-001431-12 (EudraCT Number)
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor
Keywords: TGF Beta
MeSH Terms: conditions — Camurati-Engelmann Syndrome | interventions — LY3300054; Gemcitabine; 130-nm albumin-bound paclitaxel; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- LY3200882 Schedule 1 Escalation (Experimental)
  Interventions: Drug: LY3200882
- LY3200882 Schedule 2 Escalation (Experimental)
  Interventions: Drug: LY3200882
- LY3200882 Schedule 1 Expansion (Experimental)
  Interventions: Drug: LY3200882
- LY3200882 Schedule 2 Expansion (Experimental)
  Interventions: Drug: LY3200882
- LY3200882 + LY3300054 (Experimental)
  Interventions: Drug: LY3200882; Drug: LY3300054
- LY3200882 + Gemcitabine + nab-Paclitaxel (Experimental)
  Interventions: Drug: LY3200882; Drug: Gemcitabine; Drug: nab-Paclitaxel
- LY3200882 + Cisplatin + Radiation (Experimental)
  Interventions: Drug: LY3200882; Drug: Cisplatin; Radiation: Intensity Modulated Radiotherapy
- Japanese Arm LY3200882 (Experimental)
  Interventions: Drug: LY3200882

INTERVENTIONS:
Drug: LY3200882 — Administered orally
Drug: LY3300054 — Administered intravenously
  Arms: LY3200882 + LY3300054
Drug: Gemcitabine — Administered intravenously
  Arms: LY3200882 + Gemcitabine + nab-Paclitaxel
Drug: nab-Paclitaxel — Administered intravenously
  Arms: LY3200882 + Gemcitabine + nab-Paclitaxel
Drug: Cisplatin — Administered intravenously
  Arms: LY3200882 + Cisplatin + Radiation
Radiation: Intensity Modulated Radiotherapy
  Arms: LY3200882 + Cisplatin + Radiation

SUMMARY:
The main purpose of this study is to evaluate the safety of the study drug known as LY3200882 in participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have histological or cytological evidence of cancer.
* Have adequate organ function.
* Have Eastern Cooperative Oncology Group (ECOG) scale performance status of 0 or 1.
* Are able to swallow capsules and tablets.

Exclusion Criteria:

* Have moderate or severe cardiovascular disease.
* Have a serious concomitant systemic disorder.
* Have acute leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Estimated)
Dates: Start 2016-11-21 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs) | Cycle 1 (28 days)
Part B: Overall Response Rate (ORR): Percentage of Participants with Complete Response (CR) or Partial Response (PR) | Baseline through Disease Progression or Death (estimated at up to 12 months)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Curve (AUC) (AUC[0-24]) at Steady State of LY3200882 | Cycle 1 Day 1 through Cycle 2 Day 14 (28 day cycles)
PK: AUC Zero to Infinity (AUC[0-∞]) at Steady State of LY3200882 | Cycle 1 Day 1 through Cycle 2 Day 14 (28 day cycles)
ORR: Percentage of Participants with CR or PR | Baseline through Disease Progression or Death (estimated at up to 12 months)
Overall Survival (OS) | Baseline to Date of Death from Any Cause (estimated at up to 12 months)
Duration of Response (DoR) | Date of CR or PR to Date of Disease Progression or Death Due to Any Cause (estimated at up to 12 months)
Progression-Free Survival (PFS) | Baseline to Disease Progression or Death (estimated at up to 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (18):
- United States (3):
  - University of Louisville, Louisville, Kentucky
  - Weill Cornell Medical College, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Greenslopes Private Hospital, Greenslopes, Queensland
- Princess Margaret Hospital (Ontario), Lai Chi Kok, Kowloon, Canada
- France (3):
  - Hopital Saint-Louis, Paris, Cedex 10
  - CHRU de Lille, Lille
  - Gustave Roussy, Villejuif
- Germany (2):
  - Universitätsklinikum Würzburg A. ö. R., Würzburg, Bavaria
  - Charité Campus Virchow-Klinikum, Berlin
- Italy (2):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Ospedale Policlinico Giambattista Rossi, Borgo Roma, Verona
- National Cancer Center Hospital, Chuo-Ku, Tokyo, Japan
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Yap TA, Vieito M, Baldini C, Sepulveda-Sanchez JM, Kondo S, Simonelli M, Cosman R, van der Westhuizen A, Atkinson V, Carpentier AF, Lohr M, Redman R, Mason W, Cervantes A, Le Rhun E, Ochsenreither S, Warren L, Zhao Y, Callies S, Estrem ST, Man M, Gandhi L, Avsar E, Melisi D. First-In-Human Phase I Study of a Next-Generation, Oral, TGFbeta Receptor 1 Inhibitor, LY3200882, in Patients with Advanced Cancer. Clin Cancer Res. 2021 Dec 15;27(24):6666-6676. doi: 10.1158/1078-0432.CCR-21-1504. Epub 2021 Sep 21. PMID 34548321
- See also: Click here for more information about this study: A Study of LY3200882 in Participants With Solid Tumors — http://www.lillytrialguide.com/en-US/studies/solid-tumor/JECA#?postal=